CLINICAL TRIAL: NCT00212199
Title: Effectiveness of Brief Counseling for Weight Management
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Hoffmann-La Roche (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DK58299 (completed 2205)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2010-03-18 (Estimated); Status verified 2010-03

CONDITIONS: 1. Obesity
Keywords: Obesity Treatment; Effectiveness of weight management treatment; Counseling for weight management
MeSH Terms: interventions — Orlistat

INTERVENTIONS:
Drug: orlistat
Behavioral: Brief cognitive behavioral counseling

SUMMARY:
The purpose of this study is to test the effectiveness of three different methods for delivering weight management information. Two methods utilize an obesity drug and the third method utilizes brief behavioral counseling sessions only.

DETAILED DESCRIPTION:
There is a growing demand for effective obesity treatments that don't require much time to implement especially in a primary health-care setting where time is especially limited. Brief interventions that might provide benefits similar to those produced by more time-intensive and costly lifestyle interventions would be very useful. There is also increasing interest in the efficacy of primary drug therapies for obesity. The purpose of this 12-month study, and 24-month follow-up, is to examine the efficacy of a brief behavioral counseling intervention alone or in combination with a drug already approved for the long-term management of obesity (orlisat)and compare both interventions to a drug alone condition.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index of 30 to 40
* Male or females ages of 25 to 55 years
* Normal blood pressure or controlled with medicine
* Females not lactating, able to get pregnant or using acceptable birth control
* Current allowed medications prescribed at least 2 months prior to study

Exclusion Criteria:

* Pregnant, planning to get pregnant or becomes pregnant
* Insulin dependent diabetes
* Uncontrolled hypertension
* Prescence or history of significant medical conditions that could impact the outcome of the study
* Prescence of active gastrointestinal disorders
* History of mental disorders including eating disorders
* Weight loss greater than 10 pounds in the last 3 months
* History of alcohol or drug dependency
* Use of any weight-loss medication in the last 6 months
* Known allery to orlistat or any of its components

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 246
Dates: Start 2002-01; Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
1. Changes in body weight at 6, 12 and 24 months.
2. Changes in body mass index (BMI) at 6, 12 and 24 months.

SECONDARY OUTCOMES:
1. Changes in blood pressure at 6, 12 and 24 months.
2. Changes in lipids at 6, 12 and 24 months.
3. Changes in serum glucose at 6, 12 and 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: John P Foreyt, PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States